CLINICAL TRIAL: NCT05517577
Title: Effectiveness of an Integrated Community-based Intervention Package in Improving Maternal, and Neonatal Health Outcome in Jimma Zone, Southwest Ethiopia: a Cluster Randomized Controlled Trial
Brief Title: An Integrated Community-based Intervention Package in Improving Maternal and Neonatal Health Outcomes
Acronym: ICBIP-MNH)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jimma University (Other)
Responsible Party: Principal Investigator, Bekelu Teka Worku, Lecturer and researcher, Jimma University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: JUIH/IRB/110/22
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Integrated Community-based Intervention Package; Breastfeeding, Exclusive; Morbidity;Newborn; Complementary Feeding; Knowledge, Attitudes, Practice; Food Security; Birth Preparedness and Complication Readiness Plan; Neonatal Care; Health Care Seeking Behavior; Delivery Care; Postnatal Care
Keywords: community-based intervention,; maternal,; neonatal,; infant,; health outcome,; randomized controlled trial
MeSH Terms: conditions — Breast Feeding; Behavior; Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: First, we selected two districts that have similar characteristics and are adjacent to each other. Both districts have a total of 72 kebeles (the smallest administrative unit), 36 in each district. Then, we chose 20, 10 from each district, kebeles on the boundary of the two districts to act as a buffer zone, to prevent information contamination between the intervention and control clusters. Finally, 26 kebeles in the Dedo district will be assigned to the intervention group while 26 kebeles in the Seka Chekorsa district are assigned to control clusters
Who Masked: Outcomes Assessor
Masking Description: Allocation concealment will not be done for study participants, as they would certainly know if they are in the intervention group or not. However, data collectors will be blinded to the allocation assignment by not being informed about it, not being part of the trial implementers, and not being inhabitants of any of the kebeles. Moreover, data analysts will be blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): An integrated Community-based package of interventions An integrated intervention consisting of behaviourchange communication, and male involvement will be delivered to pregnant women in their third trimester. They will receive 2 prenatal and five home visits. each visit will last 40-60 minutes. After delivery mother-newborn pairs will be followed up until six weeks.
  Interventions: Behavioral: Behaviour Change Communication and Male involvement intervention
- Control group (No Intervention): First, we selected two districts that have similar characteristics and are adjacent to each other. Both districts have a total of 72 kebeles (the smallest administrative unit), 36 in each district. Then, we chose 20, 10 from each district, kebeles on the boundary of the two districts to act as a buffer zone, to prevent information contamination between the intervention and control clusters. Finally, 26 kebeles in the Dedo district will be assigned to the intervention group while 26 kebeles in the Seka Chekorsa district are assigned to control clusters. Allocation concealment will not be done for study participants, as they would certainly know if they are in the intervention group or not. However, data collectors will be blinded to the allocation assignment by not being informed about it, not being part of the trial implementers, and not being inhabitants of any of the kebeles. Moreover, data analysts will be blinded to group allocation.

INTERVENTIONS:
Behavioral: Behaviour Change Communication and Male involvement intervention — For the integration of the intervention, it is planned to deliver both service at the same time a by the same means to the women and the men. Pregnant women who fail to take one of the intevetion will not be considered as the participant who received integrated intervention. The intervention will be provided through Women Developmental army (WDA) leaders imparted through gatherings and home visits whereas the Broadcast will be used to strengthen and as a frequent remidinng of the conveyed messages.
  Other Names: BCC
  Arms: Intervention group

SUMMARY:
This study aims to improve maternal, neonatal and infant health outcomes through an integrated community-based intervention package in Jimma Zone, Southwest Ethiopia.

DETAILED DESCRIPTION:
Background: Maternal, newborn, infant's morbidity and mortality are unacceptably high in sub-Saharan Africa including Ethiopia. Despite considerable efforts made in maternal and child health care, poor maternal, neonatal and child health problems remained a significant public health concern globally and particularly in low and middle-income countries. Community-based Interventions and strategies for improving maternal, newborn, and child health care have been recommended through a continuum of care approach. However, few efforts have been made to identify synergies and integrate different intervention packages across the country.

Objective: This study aims to assess the effectiveness of an integrated community-based intervention package in improving maternal, neonatal and infant health outcomes in Jimma Zone, Southwest Ethiopia: a cluster randomized controlled trial.

Methods: This is a parallel-arm, single-blind, cluster randomized controlled trial conducted in the Dedo and Seka Chekorsa districts of the Jimma zone. After excluding 10 kebeles from each district to be considered as a buffer zone, we will assign 26 kebeles to the intervention arm and 26 to the control arm. A total of 624 pregnant women in their third trimester who reside in the kebeles assigned to the intervention clusters will be identified and enrolled (312 in intervention and 312 in control groups). The intervention includes Behavioral Change Communication, and male involvement. Various multidisciplinary professionals and experts regularly monitor the overall process of the research and intervention activities. The effect of the intervention in comparison with the routine care will be assessed by fitting mixed-effects linear regression models for the continuous outcomes and mixed-effects linear probability models for the binary outcomes. In all analyses, adjustment will be made for clustering at the kebele level and covariate. All tests will be two-sided and the level of significance will be set at alpha < 0.05.

Budget: A total of 579,888.4ETB will be required. Key words: community-based intervention, maternal, neonatal, infant, health outcome, randomized controlled trial

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in the third trimester
* Live in the selected cluster

Exclusion Criteria:

* Serious illness or clinical complications requiring hospitalization
* Maternal death
* Newborn death
* Stillbirth
* Twin gestation
* Preterm birth (at <37 weeks)

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 624 (Estimated)
Dates: Start 2022-08-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
Neonatal care practices | At month one after delivery
  Prevalence of neonatal care practices
Feeding practice | At month one after delivery
  prevalence of early initiation and exclusive breastfeeding

SECONDARY OUTCOMES:
Neonatal morbidity | At month one after delivery
  Prevalence of neonatal morbidity
Maternal morbidity | At month one after delivery
  Prevalence of maternal morbidity
Birth preparedness and complication readiness plan | At month one after delivery
  Proportion of women who had Birth preparedness and complication readiness plan
Maternal feeding practice | : At month one after delivery
  Prevalence of minimum dietary diversity
Skilled delivery | At month one after delivery
  Prevalence of women who delivered at health institution

CONTACTS AND LOCATIONS:
Overall Officials: Bekelu Teka, MPH, Principal Investigator — Jimma University
Locations (1):
- Jimma University, Jimma, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: No